CLINICAL TRIAL: NCT03749707
Title: HPV-testing of Sentinel Lymph Node Tissue From Cervical Cancer Patients.
Brief Title: HPV in Sentinel Lymph Nodes of Cervical Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SLN2018
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-01

CONDITIONS: Cervical Cancer; Sentinel Lymph Node; HPV-Related Cervical Carcinoma
Keywords: HPV; Cervical cancer; SLN
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Early-stage cervical cancer patients treated with radical surgery and removal of SLNs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLNs from early-stage cervical cancer patients (Other): Tissue from SLNs removed from early-stage cervical cancer patients are analyzed for HPV.
  Interventions: Diagnostic Test: HPV analysis

INTERVENTIONS:
Diagnostic Test: HPV analysis — HPV analysis of SLNs with an in-house targeted Next Generation Sequencing assay

SUMMARY:
This study examines sentinel lymph node tissue from early stage cervical cancer patients treated with radical surgery and removal of pelvic sentinel lymph nodes (SLN). SLNs are tested for the presence of human papilloma virus (HPV), and results are compared to the HPV-type found in the patient's cervical tissue.

We hereby examine whether pathologic status of SLNs in patients with early-stage cervical cancer correlates to the HPV status in the SLNs. By means of an up to 5-years follow-up period, we furthermore examine whether cervical cancer recurrence correlates to the histopathologic status of the SLNs and/or the SLN HPV status. This will contribute to the clarification on whether HPV status of the SLNs plays a crucial role for predicting LN metastasis of cervical cancer and also, whether the HPV status in SLNs may have a clinical value as a prognostic factor for disease recurrence in cervical cancer patients and perhaps even a better clinical value than SLN mapping.

DETAILED DESCRIPTION:
The aim of the study is to examine whether the pathologic status of SLNs in patients with early-stage cervical cancer correlates to the HPV status in the SLNs and also, whether cervical cancer recurrence correlates to the histopathologic status of the SLNs and/or the SLN HPV status.

In Denmark, staging and treatment of cervical cancer are performed according to the recommendations of the International Federation of Gynecology and Obstetrics (FIGO). Cervical cancer is the only gynecological cancer that is clinically based on tumor size, vaginal or parametrial involvement, bladder/rectum extension and distant metastases. It requires examination under anesthesia and imaging, which in Denmark includes positron emission computed tomography (PET-CT) to detect pathological lymph nodes (LNs) and to accurately delineate the extent of the disease and magnetic resonance imaging (MRI) to determine tumor size, degree of stromal penetration, parametrial involvement, vaginal and corpus extension. Tumor risk assessment includes tumor size, stage, depth of tumor invasion, LN status, lymphovascular space invasion (LVSI) and histological subtype, of which LN status and number of LNs involved are the most important prognostic factors. In Denmark, patients at FIGO stages 1B1 to 2A undergo radical surgery and removal of SLNs, and these lymph nodes are examined by means of the ultrastaging protocol (see https://www.sciencedirect.com/science/article/pii/S0090825821005126?via%3Dihub). In this study, we want to examine the remains from these analyzed SLNs. Ultrastaging entails cutting the SLNs in more sections and all levels of the lymph node, and these levels are subsequently histologically analysed by an experienced pathologist. In this study, we examine the remains from the SLNs; that is the sections between the tissue used for SLN mapping. These sections are analyzed for HPV DNA by means of our in-house targeted Next Generation Sequencing panel (see https://febs.onlinelibrary.wiley.com/doi/10.1002/1878-0261.13538).

ELIGIBILITY:
Inclusion Criteria:

* Woman > 18 years of age diagnosed with cervical cancer and admitted for surgery with radical hysterectomy and removal of SLNs between October 2018 and June 2022.

Exclusion Criteria:

* Woman < 18 years
* Women with late-stage cervical cancer, who are treated with radio- and chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Early-stage cervical cancer patients admitted for surgery with radical surgery and removal of SLNs.
Enrollment: 127 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
HPV | 0 hours post-operation
  The presence of HPV in SLNs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Aarhus, Denmark